CLINICAL TRIAL: NCT03093311
Title: Near Infrared Spectroscopy for Detection of Cerebral Desaturation After Positioning for Neurosurgical Procedure
Brief Title: Near Infrared Spectroscopy for Detection of Cerebral Desaturation After Positioning for Neurosurgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, University Hospital Hradec Kralove, Czech Republic, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHHradecKralove 2017/01
Record Dates: First submitted 2017-03-14; First posted 2017-03-28 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Dysfunction; Patient Positioning
Keywords: Near-Infrared Spectroscopy; Neurosurgical Procedures; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Brain tissue oxygenation is measured by NIRS. In time of desaturation the interventions according to NIRS based protocol start.
  Interventions: Other: NIRS based protocol
- Arm B (No Intervention): Brain tissue oxygenation is not measured.

INTERVENTIONS:
Other: NIRS based protocol — Each desaturation episode will be managed according to a standardized protocol - correction of extreme head position will be followed by optimisation of mean arterial pressure (MAP), arterial hemoglobin oxygen saturation, end tidal carbon dioxide concentration and a level of hemoglobine concentration.
  Arms: Arm A

SUMMARY:
The occurrence of postoperative cognitive dysfunction (POCD) might be related to intraoperative cerebral desaturation. Positioning for neurosurgical procedures are associated with head rotation, elevation, flexion or extention that may affect blood brain inflow and outflow. Anatomical variations of Willis circle could affect the cerebral blood flow in extreme head position with the development of cerebral ischemia or functional changes of brain. Investigators suppose that detection of cerebral tissue desaturation and its prompt correction could modify the occurence of POCD after these procedures.

DETAILED DESCRIPTION:
Standardized anesthesia and perioperative care will be provided to all patiens with positioning for neurosurgical or spinal procedures, where the head is elevated, extended. flected or rotated. In group A before the start of general anesthesia, the baseline level of cerebral tissue oxygenation (rScO2) will be measured using the near-infrared spectroscopy NIRS (Invivo Medtronic) . Continuous measurement of rScO2 will be used for detection of cerebral tissue desaturation. Each desaturation episode will be managed according to a standardized protocol - correction of extreme head position will be followed by optimalisation of mean arterial pressure (MAP), arterial hemoglobin oxygen saturation, end tidal carbon dioxide concentration and a level of hemoglobine concentration. In group B neither measurement of rScO2 nor interventions are provided. Cognitive dysfunction will be assessed by Adenbrooke test before operation and on the fifth postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale 15, American Society of Anaesthesiologists (ASA) Physical Status Classification System Grade I-III, patient positioning with elevation, rotation, flexion or extention of head

Exclusion Criteria:

* Inability to past the Addenbrooke test, postoperative ventilation, awake phase during surgery, lung disease with retention of carbon dioxide, neurological disease before surgery (aphasia, paresis, blindness, deafness)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction of incidence of postoperative cognitive dysfunction (POCD) | 1 day before operation and the fifth´day
  Addenbrooke test

SECONDARY OUTCOMES:
Operative position of patient | first 30 minutes
  In grades from neutral position
Age of patients | the first 5 minutes
  18 to 79
Level of exhaled carbon dioxide | every 5 minutes
  In torr
Type and duration of procedure | 10 minutes after procedure
  In minutes
Dose of catecholamines | 5 minutes after procedure
  In microgramms per kg per minute

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD, PhD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No